CLINICAL TRIAL: NCT07113561
Title: Effects of a High-protein Diet and Resistance Training on Fat-mass Loss Maintenance
Acronym: PRO-FIT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: University of Alabama at Birmingham (Other); University of Leeds, Appetite Control and Energy Balance Research (Unknown); University of Copenhagen (Other); St.Olavs Hospital, Trondheim University Hospital, Norway (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 592611
Record Dates: First submitted 2025-07-08; First posted 2025-08-08 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Obesity (Body Mass Index >30 kg/m2)
MeSH Terms: conditions — Obesity | interventions — Diet, High-Protein; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-protein diet and resistance training (Experimental): Intervention group: Participants will undergo a low-calorie high-protein diet for 10 weeks, followed by a maintenance phase up to the 1-year mark. This group will also participate in supervised resistance training sessions.
  Interventions: Other: High-protein diet and resistance training
- Balanced control diet (Experimental): Control group: Participants will undergo a balanced low-calorie diet for 10 weeks, followed by a maintenance phase up to the 1-year mark. This group will not receive any active exercise intervention.
  Interventions: Other: Balanced control diet

INTERVENTIONS:
Other: High-protein diet and resistance training — Participants will consume a low-energy high-protein diet for 10 weeks, and participate in supervised resistance training sessions. They will continue a maintenance diet up until the 1 year mark, with bi-monthly follow ups on diet and exercise.
  Arms: High-protein diet and resistance training
Other: Balanced control diet — Participants will consume a balanced low-energy diet for 10 weeks, and continue a balanced maintenance diet with bi-monthly follow ups up until the 1-year mark No active exercise intervention.
  Arms: Balanced control diet

SUMMARY:
This clinical trial investigates whether a high-protein diet combined with resistance training is more effective than a standard low-calorie diet for maintaining fat mass loss in individuals with obesity.

A total of 60 adults with obesity (BMI ≥30 kg/m²) will be randomly assigned at baseline to one of two groups:

1. A control group receiving a balanced low-calorie diet.
2. An intervention group receiving a high-protein, low-calorie diet and supervised resistance training.

All participants will follow their assigned low-energy diets for the first 10 weeks, which constitutes the weight loss phase. The subsequent 42 weeks comprise the weight maintenance phase, where participants will follow an energy-balanced diet adapted to their individual needs and continue in their assigned group.

The intervention group will also complete supervised resistance training three times per week during the first 10 weeks, with continued follow-up throughout the maintenance phase.

Assessments will take place at baseline, week 11, 6 months, and 12 months, and include measurements of fat and lean mass, resting metabolic rate, appetite hormones, glucose metabolism, inflammation, gut microbiota and its metabolites, hedonic appetite, eating behavior, and quality of life and physical function. Participants will also provide food intake records, physical activity dat.

The primary aim is to determine whether the combined high-protein diet and resistance training intervention results in greater long-term fat mass loss and muscle mass preservation than the control diet. Secondary aims include effects on appetite regulation, eating behavior, metabolic health, and patient-reported outcomes.

The study is conducted at NTNU and St. Olavs Hospital in Trondheim, Norway, and registered under the acronym PRO-FIT.

ELIGIBILITY:
Inclusion Criteria:

* BMI equal to or above 30
* Sedentary lifestyle (<150 minutes moderate physical activity per week and no habitual resistance training (< once weekly)
* < 2 kg body weight change in the 3 months prior to study commencement
* high motivation for lifestyle change
* not currently enrolled in any other obesity or behavioral change program

Exclusion Criteria:

* Previous or planned bariatric surgery
* Current or planned usage of medications or anti-obesity drugs known to influence energy metabolism or appetite
* Diabetes (type 1 and 2)
* Women in menopause or post-menopausal women
* Existing cancer diagnosis
* Renal disease
* Substance abuse
* Eating disorders
* Allergies, or intolerances to ingredients in meal packs/supplements intended for use in the study
* Mobility/physical constrains or musculoskeletal issues that could impede participation in the resistance training program

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Fat-mass | From enrollment at baseline , after 10 weeks of weight loss phase, and at 52 weeks.
  Fat-mass will be estimated using a dual-energy absorptiometry (DXA, GE Healthcare Lunar).
Fat-free mass | From enrollment at baseline , after 10 weeks of weight loss phase, and at 52 weeks.
  Fat-free mass will be estimated using a dual-energy absorptiometry (DXA, GE Healthcare Lunar).

SECONDARY OUTCOMES:
Body weight and -composition | From enrollment at baseline , after 10 weeks of weight loss phase, 26 and at 52 weeks.
  Body weight and -composition will be estimated with dual-energy absorptiometry (DXA, GE Healthcare Lunar) (primary outcomes) and bioimpedance (InBody 770). Compartments that will be estimated are: total body weight, Fat-mass, fat-free mass, bone mineral density, visceral fat, muscle mass, body water, as well as segmental analysis of body weight and composition.
Anthropometric variables | From enrollment at baseline , after 10 weeks of weight loss phase, 26 and at 52 weeks.
  Height, hip- and waist circumference will be measured using standardized methods. Body weight and height will be used to calculate body mass index in kg/m^2. Hip-, waist- and height measurements will be used to calculate height/waist- and hip/waist ratio.
Resting metabolic rate | From enrollment at baseline , after 10 weeks of weight loss phase, and at 52 weeks.
  Resting metabolic rate will be measured in the fasted state using an indirect calorimetry (Quark RMR, Cosmed).
Leeds food preference questionnaire | From enrollment at baseline , after 10 weeks of weight loss phase, and at 52 weeks.
  Food reward and -preferences will be assessed with the Leeds Food Preference Questionnaire (LFPQ), in the fasted state and immediately after the test meal. The LFPQ is a computerized behavioral task that provides measures of 'explicit liking' and explicit and 'implicit wanting' for sensory and nutrient dimensions of foods using food images.
Dutch Eating Behavior Questionnaire | From enrollment at baseline , after 10 weeks of weight loss phase, and at 26 and 52 weeks.
  The Dutch Eating Behavior Questionnaire measures restrained, external and emotional eating. Emotional eating can be divided into two sub-categories: diffuse emotions and clearly labelled emotions. The greater score, the greater external/emotional eating.
Power of Food Scale | From enrollment at baseline , after 10 weeks of weight loss phase, and at 26 and 52 weeks.
  The Power of food scale is a psychometric evaluation that measures an individual's preoccupation with wanting of highly palatable foods. The PFS consists of a 15-item list that measures hedonic hunger (food-related thoughts that are unrelated to homeostatic need). The higher the PFS score, the greater the hedonic hunger.
Three Factor Eating Questionnaire | From enrollment at baseline , after 10 weeks of weight loss phase, and at 26 and 52 weeks.
  The Three Factor Eating Questionnaire measures three different dimensions: restraint, disinhibition, and hunger. The greater score, the stronger is the trait/behavior.
Ghrelin | From enrollment at baseline , after 10 weeks of weight loss phase, and at 52 weeks.
  Blood will be collected in the fasted state (minute 0), and then at intervals after a standardized breakfast (minute 15, 30, 45, 60, 90, 120 and 150) and analyzed for acylated ghrelin concentrations.
GLP-1 | From enrollment at baseline , after 10 weeks of weight loss phase, and at 52 weeks.
  Blood will be collected in the fasted state (minute 0), and then at intervals after a standardized breakfast (minute 15, 30, 45, 60, 90, 120 and 150) and analyzed for total GLP-1 concentrations.
CCK | From enrollment at baseline , after 10 weeks of weight loss phase, and at 52 weeks.
  Blood will be collected in the fasted state (minute 0), and then at intervals after a standardized breakfast (minute 15, 30, 45, 60, 90, 120 and 150) and analyzed for CCK concentrations.
PYY | From enrollment at baseline , after 10 weeks of weight loss phase, and at 52 weeks.
  Blood will be collected in the fasted state (minute 0), and then at intervals after a standardized breakfast (minute 15, 30, 45, 60, 90, 120 and 150) and analyzed for total PYY concentrations.
Insulin | From enrollment at baseline , after 10 weeks of weight loss phase, and at 52 weeks.
  Blood will be collected in the fasted state (minute 0), and then at intervals after a standardized breakfast (minute 15, 30, 45, 60, 90, 120 and 150) and analyzed for insulin concentrations.
C-peptide | From enrollment at baseline , after 10 weeks of weight loss phase, and at 52 weeks.
  Blood will be collected in the fasted state (minute 0), and then at intervals after a standardized breakfast (minute 15, 30, 45, 60, 90, 120 and 150) and analyzed for c-peptide concentrations.
Glucose | From enrollment at baseline , after 10 weeks of weight loss phase, and at 52 weeks.
  Blood will be collected in the fasted state (minute 0), and then at intervals after a standardized breakfast (minute 15, 30, 45, 60, 90, 120 and 150) and analyzed for glucose concentrations.
GIP | From enrollment at baseline , after 10 weeks of weight loss phase, and at 52 weeks.
  Blood will be collected in the fasted state (minute 0), and then at intervals after a standardized breakfast (minute 15, 30, 45, 60, 90, 120 and 150). Plasma samples will be stored and analyzed for GIP concentrations depending on additional funding.
Glucagon | From enrollment at baseline , after 10 weeks of weight loss phase, and at 52 weeks.
  Blood will be collected in the fasted state (minute 0), and then at intervals after a standardized breakfast (minute 15, 30, 45, 60, 90, 120 and 150). Plasma samples will be stored and analyzed for glucagon concentrations depending on additional funding.
IL-6 | From enrollment at baseline , after 10 weeks of weight loss phase, and at 52 weeks.
  Blood will be collected and plasma samples will be stored and analyzed for IL-6 concentrations depending on additional funding.
TNF-alfa | From enrollment at baseline , after 10 weeks of weight loss phase, and at 52 weeks.
  Blood will be collected and plasma samples will be stored and analyzed for TNF-alfa concentrations depending on additional funding.
CRP | From enrollment at baseline , after 10 weeks of weight loss phase, and at 52 weeks.
  Blood will be collected in the fasted state (minute 0), and analyzed for CRP.
Triglycerides | From enrollment at baseline , after 10 weeks of weight loss phase, and at 52 weeks.
  Blood will be collected in the fasted state (minute 0), and analyzed for triglycerides.
HbA1C | From enrollment at baseline , after 10 weeks of weight loss phase, and at 52 weeks.
  Blood will be collected in the fasted state (minute 0), and analyzed for HbA1C
HDL | From enrollment at baseline , after 10 weeks of weight loss phase, and at 52 weeks.
  Blood will be collected in the fasted state (minute 0), and analyzed for high-density lipoprotein
LDL | From enrollment at baseline , after 10 weeks of weight loss phase, and at 52 weeks.
  Blood will be collected in the fasted state (minute 0), and analyzed for low-density lipoprotein
Total cholesterol | From enrollment at baseline , after 10 weeks of weight loss phase, and at 52 weeks.
  Blood will be collected in the fasted state (minute 0), and analyzed for total choesterol.
Hemoglobin | From enrollment at baseline , after 10 weeks of weight loss phase, and at 52 weeks.
  Blood will be collected in the fasted state (minute 0), and analyzed for hemoglobin.
Gut microbiota | From enrollment at baseline , after 10 weeks of weight loss phase, and at 52 weeks.
  Fecal samples will be collected and comprehensive microbiota profiling using DNA-based sequencing will be performed.
Short-chain fatty-acids | From enrollment at baseline , after 10 weeks of weight loss phase, and at 52 weeks.
  Fecal samples will be collected and acetate, propionate, and butyrate will be quantified by gas chromatography-mass spectrometry (GC-MS)
IWQOL-lite | From enrollment at baseline , after 10 weeks of weight loss phase, and at 52 weeks.
  The Impact of Weight on Quality of Life (IWQOL)-Lite questionnaire will be used to assess obesity-specific quality of life and includes 5 subcategories: physical function, self-compassion, sexual life, public distress and work. In addition, the total quality of life score will be assessed. Higher score, better quality of life.
Short Form-36 (SF-36) | From enrollment at baseline , after 10 weeks of weight loss phase, and at 52 weeks.
  The SF-36, or Short Form 36, is a 36-item questionnaire used to assess a person's self-reported health-related quality of life. It measures eight health concepts: physical functioning, role limitations due to physical health, bodily pain, general health, vitality, social functioning, role limitations due to emotional health, and mental health where a higher score represents better health.
Estimated one-repetition maximum (1RM) | From enrollment at baseline , after 10 weeks of weight loss phase, and at 26- and 52 weeks.
  1RM will be calculated using submaximal lifts performed to muscular failure within 4-8 repetitions.
Patient specific functional Scale | From enrollment at baseline , after 10 weeks of weight loss phase, and at 52 weeks.
  The Patient Specific Functional Scale is a patient-specific instrument. This means that the patient selects activities (three to five) that they have difficulty performing due to their illness or injury, and then rates their ability to perform these activities.
Force development- and peak force | From enrollment at baseline , after 10 weeks of weight loss phase, and at 52 weeks.
  A one-repetition max tests and a force development- and peak force task will be undertaken on a force platform (Kistler, Switzerland) installed on a leg press device.
Subjective appetite | From enrollment at baseline , after 10 weeks of weight loss phase, and at 52 weeks.
  Subjective ratings of appetite (hunger, fullness, desire to eat, and prospective food consumption) will be measured in fasting (minute 0) and then at minute 15, 30, 60, 90, 120 and 150 after the standardized test meal.
Blood pressure | From enrollment at baseline , after 10 weeks of weight loss phase, and at 52 weeks.
  Blood pressure will be measured in units of millimeters of mercury (mmHg)

OTHER OUTCOMES:
Food records | Before start of intervention, during weight loss phase, at 6 month follow up, and prior to assessments at week 52.
  Participants will quantify their daily energy intake by logging self-reported food diaries. Energy intake and macronutrient distribution will be calculated based on reported foods and quantitates.
Ketone bodies | At baseline assessments, during weight loss phase( baseline to week 11), at week 11 assessments, at 6 months and assessments at week 52
  In addition to food logs, ketone bodies will be measured for compliance to diet and to account for potential nutritional induced ketosis. Acetoacetate will be measured in urine using Bayer ketostix and betahydroxtbutyrate using a freestyle libre ketone meter.
Plasma samples | From enrollment at baseline , after 10 weeks of weight loss phase, and at 52 weeks.
  Plasma samples will also be stored for exploratory analyses later
Adherence to exercise intervention | During weight loss phase( baseline to week 11), and during maintenance phase up until week 52
  Attendance to scheduled training sessions will be recorded, together with type of exercise, sets, reps and loads.
Physical activity levels | Before and during weight loss phase( baseline to week 11), at 26 and 52 weeks
  Physical activity levels will be estimated using actigraphs for 7-day periods.

CONTACTS AND LOCATIONS:
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided